CLINICAL TRIAL: NCT07202156
Title: Clinical Trial on the Efficacy and Safety of Ultrasound-Enhanced Delivery of Compound Tranexamic Acid Solution in the Treatment of Melasma
Brief Title: Ultrasound-Enhanced Delivery of Compound TXA Solution in Melasma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR-820
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Melasma (Facial Melasma)
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical treatment with Ultrasound (Experimental): 10%TXA+2%Reduced Glutathione applied via ultrasound at 5W/cm² for 10mins
  Interventions: Device: 10%TXA+2%Reduced Glutathione applied via ultrasound at 5W/cm² in10min
- Topical treatment without Ultrasound (Other): 10%TXA+2%Reduced Glutathione applied via ultrasound at 0W/cm² for 10mins
  Interventions: Other: 10%TXA+2%Reduced Glutathione applied via ultrasound at 0W/cm² 10min

INTERVENTIONS:
Device: 10%TXA+2%Reduced Glutathione applied via ultrasound at 5W/cm² in10min — 5w/cm² Ultrasound-assisted topical application of 10% tranexamic acid and 2% reduced glutathione for 10 mins
  Arms: Topical treatment with Ultrasound
Other: 10%TXA+2%Reduced Glutathione applied via ultrasound at 0W/cm² 10min — topical application of 10% tranexamic acid and 2% reduced glutathione for 10 mins
  Arms: Topical treatment without Ultrasound

SUMMARY:
Melasma is a localized, acquired hyperpigmentary skin disorder characterized by well-defined, light to dark brown patches. Based on clinical practice and extensive literature reports, tranexamic acid and reduced Glutathione (GSH) are both applied in the treatment of melasma, but their water-soluble nature presents challenges for transdermal absorption. Our preliminary basic and clinical research has demonstrated that ultrasound-assisted delivery significantly enhances the absorption of tranexamic acid and other water-soluble components. Its effect on the skin barrier is temporary and reversible.

This study aims to evaluate the efficacy and safety of a compound solution (10% tranexamic acid, 2% GSH) delivered via ultrasound for melasma treatment through a split-face controlled trial.

ELIGIBILITY:
Inclusion Criteria:

-(1) Male or female participants aged 20 to 55 years (inclusive); (2) Subjects clinically diagnosed with melasma and confirmed by the investigator to meet the trial requirements; (3) Subjects willing to comply with follow-up observations and able to provide portrait rights for documentation purposes; (4) Understanding and willingness to participate in the clinical trial, and voluntarily signing a written informed consent form.

Exclusion Criteria:

* (1) Females who are pregnant, lactating, or planning to become pregnant during the trial period; (2) Subjects with known allergen to tranexamic acid or any excipient in the investigational product; (3) History of thrombosis or other thrombotic tendencies (e.g., hypertension, hyperlipidemia), or inability to discontinue oral contraceptives, estrogen, or prothrombin complex concentrates during the trial; (4) History of visual or ocular abnormalities (e.g. impaired vision, visual field defects, or fundus hemorrhage/edema) caused by abnormal retinal intravascular coagulation; (5) Patients with skin inflammation who have used topical steroid preparations for more than one month; (6) Presence of skin abnormalities at the trial site, such as nevi, ulcers, or erosions; (7) Any acute or chronic medical history (past or present) that may interfere with the validity or safety assessment of the trial; (8) Clinically significant abnormal laboratory test results prior to the trial; (9) Participation in any other clinical trial within 30 days prior to screening; (10) Any other condition deemed by the investigator to be unsuitable for participation in the study.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
percentage reduction in hemi-MASI | From enrollment to the end of treatment at 8 weeks, and 4&12 weeks after the final intervention
  mean percentage reduction in hemi-MASI from baseline to week 20

SECONDARY OUTCOMES:
Patient self-assessment | week 4 during treatment and the end of treatment at 8 weeks, and 4&12 weeks after the final intervention
  The outcomes were categorized as follows: cured (improvement ≥75%), markedly effective (improvement 50%-75%), effective (improvement 25%-50%), and ineffective (improvement ≤25%). The satisfaction rate was calculated as: Satisfaction rate = (number of cured + markedly effective + effective cases) / total number of cases × 100%
Clinical Efficacy | week 4 during treatment and the end of treatment at 8 weeks, and 4&12 weeks after the final intervention
  investigators evaluated the melasma or hyperpigmentation on split-face using the following criteria: Cured: >90% reduction in pigmented area with virtually disappearance of color upon visual inspection.
  Markedly Effective: >60% reduction in area with significant lightening of color.
  Effective: >30% reduction in area with noticeable lightening of color. Ineffective: <30% reduction in area with no significant change in color. The effective rate was calculated as: Effective rate = (number of cured + markedly effective + effective cases) / total number of cases × 100%.
VISIA Digital Skin Analysis | From enrollment to the end of treatment at 8 weeks, and 4&12 weeks after the final intervention
Melasma Quality of Life Scale (MELASQOL) Score | The enrollment, week 4 during treatment and the end of treatment at 8 weeks, and 4&12 weeks after the final intervention

OTHER OUTCOMES:
Two-Photon Microscopic Imaging | The enrollment, week 4 during treatment and the end of treatment at 8 weeks, and 4&12 weeks after the final intervention
  This was to monitor experimental safety and the impact on the skin barrier.
Dermatoscopy | The enrollment, week 4 during treatment and the end of treatment at 8 weeks, and 4&12 weeks after the final intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lu Yan, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first Affiliated hospital with Nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No